CLINICAL TRIAL: NCT00407355
Title: A Pilot, Open-Label Study of the Safety, Tolerability, and Bioactivity of Multiple Intravitreal Injections of Ranibizumab in Subjects With Macular Edema Secondary to Vein Occlusions.
Brief Title: Ranibizumab (Lucentis) for Macular Edema Secondary to Vein Occlusions
Acronym: LVO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter A Campochiaro, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Peter A Campochiaro, MD, Principal Investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-06-09-05
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: vein occlusion; macular edema
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RBZ 0.3 (Active Comparator): RBZ at the 0.3 mg dose intravitreal injection
  Interventions: Drug: Intravitreal injection of ranibizumab .3 dose
- RBZ 0.5 (Active Comparator): RBZ dose level .5 for ITV injection
  Interventions: Drug: Intravitreal injection of Ranibizumab .5 dose

INTERVENTIONS:
Drug: Intravitreal injection of ranibizumab .3 dose — PRN every 30 days withing retreatment criteria
  Arms: RBZ 0.3
Drug: Intravitreal injection of Ranibizumab .5 dose — Intravitreal injection of Ranibizumab .5 dose every 30 days PRN with retreatment criteria
  Arms: RBZ 0.5

SUMMARY:
Central and branch retinal vein occlusions are major causes of visual loss. Hemorrhage and capillary nonperfusion, when they involve the macula, can contribute to visual loss, but the major cause is macular edema. Focal and grid laser photocoagulation can sometimes provide benefit in patients with macular edema due to branch vein occlusions, but several laser treatments are often needed and recovery of vision can be very slow and incomplete 1. Laser photocoagulation does not provide benefit for macular edema due to central vein occlusions 2. Therefore, new treatments are needed.The objective of this study is to assess the bioactivity of 3 intravitreous injections 0.5 mg or 0.3 mg of ranibizumab in patients with macular edema due to central and branch retinal vein occlusions and correlate activity with peak and trough aqueous levels. The purpose of this research protocol is pilot study to determine if a randomized placebo controlled trial is warranted.

DETAILED DESCRIPTION:
This study is a phase II, open-label study to investigate the bioactivity and pharmacodynamics of intravitreous ranibizumab in subjects with macular edema due to central and branch retinal vein occlusion. This pilot study will enroll 40 patients, 20 with central vein occlusion and 20 with branch vein occlusion. Each patient will receive three (3) injections of 0.5 or 0.3 mg of ranibizumab. The study consists of a 2-week screening period (Days -14 to -1), a 3-month treatment period, and a 9-month follow-up period. Consented subjects will enter the 14-day screening period to determine eligibility, including serum chemistry and hematology testing, urinalysis, pregnancy testing, and macular thickness based on optical coherence tomography measurements and fluorescein angiography. Patients who have reduction of visual acuity to 20/40 or worse due to foveal thickening from macular edema secondary to central or branch retinal vein occlusion and who meet eligibility criteria will be invited to enroll in the study. Baseline foveal thickness by OCT must be at least 250 um, which is often associated with VA of 20/40 or worse and provides sufficient thickening so that a treatment effect is easily detectable (Nguyen et al. 2004). Every effort will be made to recruit and enroll eligible patients from men and women of all ethnic and social backgrounds. It is expected that the 40 study subjects will be recruited over a 4-month period. Patients who meet entry criteria will be able to enroll in the study until the quota of patients has been achieved. All enrolled patients will receive either 0.5 or 0.3 mg injections of ranibizumab. Forty eligible subjects who have provided informed consent from one site (Wilmer Eye Institute at the Johns Hopkins Medical Institutions) will be enrolled, 20 with central vein occlusion and 20 with branch vein occlusion. In each of the 2 groups, 10 patients will be randomized to 0.5 mg of the ranibizumab, and 10 will be randomized to 0.3 mg of ranibizumab. Subjects will be identified and recruited through the clinic population of the Wilmer Eye Institute, including that of the Vitreoretinal Service and the Retinal Vascular Center, as well as through referral from physicians in the community. Announcement of the study will be made throughout the Wilmer Eye Institute, Johns Hopkins University School of Medicine through newsletters, pamphlets, and the clinical trials web site on the internet and intranet systems. Information about the study will also be sent to the community physicians as well as the ophthalmologists who often refer patients to the Wilmer Eye Institute. Every effort will be made to enroll eligible patients from men and women of all ethnic and social backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age greater than or equal to 18 years
* Diagnosis of macular edema due to central or branch retinal vein occlusion
* Foveal thickness of over 250 um, as assessed by OCT
* Best corrected visual acuity score in the study eye of 20/40 to 20/320 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters). Only one eye will be treated in the study. If both eyes are eligible, the investigator will select the eye to be enrolled. Visual acuity score in the non-study eye must be greater than 25 letters (approximate Snellen equivalent 20/320).
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from vein occlusion and not from other obvious causes of decreased vision
* In the opinion of the investigator, laser photocoagulation can be withheld for at least 30 days after the patient has enrolled in the study

Exclusion Criteria:

* Prior/Concomitant Treatment

  * Scatter laser photocoagulation or macular photocoagulation within 3 months of study entry in the study eye
  * Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 3 months of study entry
  * Previous participation in a study and receipt of anti-angiogenic drugs (pegaptanib sodium [EYE001], ranibizumab, anecortave acetate, protein kinase C inhibitor, etc.) within 3 months of study entry Concurrent Ocular Conditions
  * Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
  * Ocular inflammation (including 1+ or above in the amount of cells) in the study eye
  * History of idiopathic or autoimmune uveitis in either eye
  * Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), macular ischemia, or organized hard exudate plaque
  * Ocular disorders in the study eye that may confound interpretation of study results, including diabetic retinopathy, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., AMD, ocular histoplasmosis, or pathologic myopia)
  * Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
  * Intraocular surgery in the study eye within 3 months of study entry
  * During the study, if patients need to have cataract surgery, the patients will undergo the necessary cataract or any other surgery and will continued to be treated per protocol and followed.
  * Uncontrolled glaucoma (defined as intraocular pressure greater than 30 mm Hg despite treatment with anti-glaucoma medication) or previous filtration surgery in the study eye
  * Infectious blepharitis, keratitis, scleritis, or conjunctivitis (in either eye) or current treatment for serious systemic infection Systemic Conditions
  * Blood pressure exceeding 160/95 (sitting) during the screening period
  * Renal failure requiring dialysis or renal transplant
  * Premenopausal women not using adequate contraception
  * Previous participation in other studies of investigational drugs (excluding vitamins and minerals) within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sophie R, Hafiz G, Scott AW, Zimmer-Galler I, Nguyen QD, Ying H, Do DV, Solomon S, Sodhi A, Gehlbach P, Duh E, Baranano D, Campochiaro PA. Long-term outcomes in ranibizumab-treated patients with retinal vein occlusion; the role of progression of retinal nonperfusion. Am J Ophthalmol. 2013 Oct;156(4):693-705. doi: 10.1016/j.ajo.2013.05.039. PMID 24053892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients with central retinal vein occlusion(CRVO) and 20 patients with branch retinal vein occlusion (BRVO) were enrolled at the Wilmer Eye Institute
Groups:
- CRVO; BRVO: 10 patients- RBZ dose level .5 for ITV injection given monthly for 3 months, then prn until 6 years 10 patients- RBZ dose level .3 for ITV injection given monthly for 3 months, then .5 prn until 6 years
Period: Overall Study
Arm/Group | CRVO | BRVO
Started | 20 | 20
Completed | 10 | 9
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRVO | BRVO | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 63.9 (15.7) | 67.4 (11.3) | 67.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity Change From Baseline at All Visits
Time Frame: continuous through 72 mos
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | CRVO | BRVO
Number analyzed (Participants) | 10 | 9
ETDRS letters | 10.5 (9.3) | 15.1 (10.7)

2. Primary Outcome: Retinal Thickness Change From Baseline at All Visits
Time Frame: continuous through 72 mos
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | CRVO | BRVO
Number analyzed (Participants) | 10 | 9
microns | -379.9 (239.1) | -216.9 (147.1)

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | CRVO | BRVO
Serious Adverse Events (participants affected / at risk) | 8/20 | 6/20
Other Adverse Events (participants affected / at risk) | 8/20 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO (N=20) | BRVO (N=20)
Vitrectomy (Eye disorders) | 1 (1) | 0 (0) — Vitrectomy done due to recurrent vitreous hemorrhage in patient.
Transient Ischemic attack (Cardiac disorders) | 1 (1) | 0 (0) — Patient admitted to hospital, diagnosed with TIA and recovered
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve surgery (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia requiring hospitalization (Infections and infestations) | 1 (1) | 1 (1)
Surgerical resection of breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Surgical resection of meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign pancreatic mass surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Scheduled surgery for hearing problem (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Death (cause unknown) (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) — Patient had pulmonary embolism following hip surgery and passed away.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO (N=20) | BRVO (N=20)
Respiratory Infection (Infections and infestations) | 8 (10) | 4 (7) — This includes, common cold, sinus infections and bronchitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No